CLINICAL TRIAL: NCT06381154
Title: Photodynamic Priming to Facilitate Immunologic Activity of Anti-PD1 in Patients With Pancreatic Cancer
Brief Title: Photoradiation With Verteporfin to Facilitate Immunologic Activity of Pembrolizumab in Unresectable, Locally Advanced or Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230404; NCI-2024-03078 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-009036 (Other: Mayo Clinic Institutional Review Board); MC230404 (Other: Mayo Clinic); P01CA084203 (NIH)
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; Specimen Handling; Endoscopic Ultrasound-Guided Fine Needle Aspiration; Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Sentinel Lymph Node Biopsy; Magnetic Resonance Spectroscopy; Oxaliplatin; pembrolizumab; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (verteportin, photoradiation, pembrolizumab) (Experimental): Patients receive verteporfin IV and undergo a biopsy and intratumoral photoradiation over 60-90 minutes using EUS or CT guidance on day 0. Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care oxaliplatin IV over 2-6 hours, leucovorin IV over 15 minutes - 2 hours, irinotecan IV over 90 minutes, and fluorouracil IV on days 3, 15 and 29 of cycle 1 only, then on days 1, 15, and 29 of remaining cycles. Cycles repeat every 42 days for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients may optionally undergo lymph node biopsy on day 2 or 3 of cycle 1. Additionally, patients undergo blood sample collection, CT, PET/CT and optional PET/MRI on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Endoscopic Ultrasound; Drug: Fluorouracil; Drug: Irinotecan; Drug: Leucovorin; Procedure: Lymph Node Biopsy; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Biological: Pembrolizumab; Drug: Photodynamic Therapy; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Verteporfin

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Endoscopic Ultrasound — Undergo EUS
  Other Names: endosonography; EUS
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan — Given IV
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Procedure: Lymph Node Biopsy — Undergo lymph node biopsy
  Other Names: Biopsy of Lymph Node
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669; Elplat; JM83; RP54780; SR96669
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475; MK3475; GME751; GME 751; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27
Drug: Photodynamic Therapy — Undergo intratumoral photoradiation
  Other Names: PDT; Photoradiation Therapy
Procedure: Positron Emission Tomography — Undergo PET/CT and PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Drug: Verteporfin — Given IV
  Other Names: Benzoporphyrin Derivative Monoacid Ring A; BPD-MA; Visudyne

SUMMARY:
This phase II trial tests how well photoradiation with verteporfin and pembrolizumab plus standard of care chemotherapy works in treating patients with pancreatic cancer that cannot be removed by surgery (unresectable), that has spread to nearby tissue or lymph nodes (locally advanced) or to other places in the body (metastatic). Photoradiation uses light activated drugs, such as verteporfin, that become active when exposed to light. These activated drugs may kill tumor cells. Vertoporfin may also increase tumor response to immunotherapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as modified fluorouracil, leucovorin, irinotecan, and oxaliplatin (mFOLFIRINOX), work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Photoradiation with verteporfin and pembrolizumab plus standard of care chemotherapy may kill more tumor cells in patients with unresectable, locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate overall response rate (ORR) per immune-mediated Response Evaluation Criteria in Solid Tumors (iRECIST) criteria in pancreatic cancer patients treated with the combination photodynamic priming (PDP) and pembrolizumab.

SECONDARY OBJECTIVES:

I. To evaluate ORR by 1st vs. 2nd line therapy. II. To evaluate duration of response (DOR) per iRECIST criteria in patients treated with the combination of PDP and pembrolizumab.

III. To evaluate progression-free survival (PFS) per iRECIST criteria in patients treated with the combination of PDP and pembrolizumab.

IV. To evaluate overall survival (OS) in patients treated with the combination of PDP and pembrolizumab.

V. To evaluate toxicity profile per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 as assessed by treating clinicians of the combination of PDP and pembrolizumab.

OTHER OBJECTIVES:

I. To evaluate the local and systemic immune response by evaluation of tumor directed cytotoxic lymphocytes within the primary and metastatic tumor sites using endoscopic ultrasound (EUS) guided fine needle aspiration before and after PDP.

II. To evaluate the biomarkers generated by the lymphocyte cytotoxicity assays using harvested lymphocytes from these sites.

III. To evaluate systemically circulating tumor directed cytotoxic lymphocyte sub-populations before and after PDP.

IV. To evaluate quality of life using Quality of Life Questionnaire-Pancreatic Cancer 26 (QLQ PAN26), European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30).

OUTLINE:

Patients receive verteporfin intravenously (IV) and undergo a biopsy and intratumoral photoradiation over 60-90 minutes using EUS or computed tomography (CT) guidance on day 0. Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care oxaliplatin IV over 2-6 hours, leucovorin IV over 15 minutes - 2 hours, irinotecan IV over 90 minutes, and fluorouracil IV on days 3, 15 and 29 of cycle 1 only, then on days 1, 15, and 29 of remaining cycles. Cycles repeat every 42 days for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients may optionally undergo lymph node biopsy on day 2 or 3 of cycle 1. Additionally, patients undergo blood sample collection, CT, positron emission tomography (PET)/CT and optional PET/magnetic resonance imaging (MRI) on study.

After completion of study treatment, patients are followed up at 30 and 90 days and every 3 months to progression then every 6 months for up to 3 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary tumor histologically or cytologically confirmed (previously biopsied) meta-static, unresectable, or locally advanced pancreatic ductal adenocarcinoma (PDAC), including malignant transformation of a mucinous tumor [intraductal papillary-mucinous neoplasm (IPMN) or mucinous cystic neoplasm (MCN)]

  * NOTE: Primary tumor in pancreas must still be present to be eligible.
* Prior treatment for this pancreatic tumor is allowed as follows:

  * Up to one line (≤1 regimen) of prior therapy is allowed
  * No prior treatment with FOLFIRINOX
* Measurable disease as defined by iRECIST. NOTE: Tumor lesions in previously irradiated area are considered measurable if previous evidence of progression has been found in these lesions
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 15 days prior to registration)
* White blood cell (WBC) ≥ 2500/mm^3 (obtained ≤ 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 15 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 15 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN ( ≥ 5 x ULN for patients with liver involvement) (obtained ≤ 15 days prior to registration)
* Prothrombin time (PT) / international normalized ratio (INR) / activated partial thromboplastin time (aPTT) ≤ x ULN (obtained ≤ 15 days prior to registration) OR if patient is receiving anticoagulant therapy then INR or aPTT is within target range of therapy
* Creatinine ≤ 1.5 x ULN (obtained ≤ 15 days prior to registration) OR calculated creatinine clearance ≥ 50 ml/min using the Cockcroft-Gault formula
* Negative pregnancy test done ≤ 8 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
* Histology or cytology of pancreatic tumor other than adenocarcinoma
* Prior treatment:

  * Received more than one regimen of treatment for pancreatic cancer
  * Received prior treatment with FOLFIRINOX
* History of immunodeficiency illness or immune suppressive medication including systemic steroid therapy or any other form of immunosuppressive therapy ≤ 7 days prior to registration
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment.

  * EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known history of human immunodeficiency virus (HIV) infection
* Concurrent active hepatitis B (defined as hepatitis B surface antigen [HBsAg] positive and/or detectable hepatitis B virus [HBV] deoxyribonucleic acid [DNA]) and hepatitis C virus (defined as anti-hepatitis C virus [HCV] antibody [Ab] positive and detectable HCV ribonucleic acid [RNA]) infection

  * EXCEPTIONS:

    * For patients with evidence of hepatitis B virus (HBV) infection (HBsAg positive), patients must have completed at least 4 weeks of HBV antiviral therapy and the HBV viral load must be undetectable at the time of registration
    * Patients with a history of hepatitis C virus (HCV) are eligible if they have an undetectable HCV viral load. Patients must have completed curative anti-viral treatment ≥ 4 weeks prior to registration
    * NOTE: Patients without symptoms or prior history do not require testing prior to registration
* History of unstable angina, new onset angina ≤ 3 months prior to registration, myocardial infarction ≤ 6 months prior to registration, or current congestive heart failure New York Heart Association class III or higher
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Current diagnosis or previous history of immune-related (non-infectious) pneumonitis or interstitial lung disease that requires or required steroids
  * Active autoimmune disease that has required systemic treatment ≤ 2 years prior to registration (i.e., with the use of disease-modifying agents, cortico-steroids, or immunosuppressive drugs) NOTE: Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy) is allowed
  * Any condition requiring systemic treatment with either corticosteroids ( > 10 mg daily prednisone equivalents) or other immunosuppressive medications. NOTE: Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Other active concurrent malignancy

  * EXCEPTIONS: Non-melanotic skin cancer, carcinoma-in-situ of the cervix, papillary thyroid cancer, or other in situ cancer that has undergone potentially curative therapy
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2029-12-06 (Estimated); Study Completion 2029-12-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of patients who achieve complete response (CR) or partial response (PR) per immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST) during protocol treatment among evaluable patients.

SECONDARY OUTCOMES:
ORR by 1st versus 2nd line therapy | Up to 2 years
  ORR will be reported separately for 1st versus 2nd line therapy groups.
Duration of response (DOR) | Up to 5 years
  DOR is defined as the time from the date of first documented CR or PR to the date of first documented disease progression per iRECIST or death due to all causes, whichever occurs first.
Progression-free survival (PFS) | Up to 5 years
  PFS is defined as the time from the date of registration to the date of first documented disease progression per iRECIST or death due to all causes, whichever occurs first.
Overall survival (OS) | Up to 5 years
  OS is defined as the time from the date of registration to the date of death due to all causes, whichever occurs first.
Incidence of adverse events (AEs) | Up to 90 days after last dose of study drug (treatment cycles are usually 29 days)
  AEs will be graded using the Common Terminology Criteria for Adverse Events version 5.0. AEs and the maximum grade for each type of AE will be summarized for each patient. Frequency tables will be reviewed to determine patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials